CLINICAL TRIAL: NCT01701635
Title: A Bioecological Pediatric HIV Disclosure Intervention in Ghana - "SANKOFA"
Brief Title: SANKOFA Pediatric HIV Disclosure Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Purdue University (Other); University of Ghana (Other); Kwame Nkrumah University of Science and Technology (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1205010310; NIH/NICHD (Other Grant/Funding Number: NIH/NICHD 074253); R01HD074253 (NIH)
Record Dates: First submitted 2012-10-02; First posted 2012-10-05 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: HIV
Keywords: Disclosure; HIV-infected children; Resource-limited settings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Disclosure intervention (Experimental): In the disclosure intervention plus usual care arm the adherence and disclosure specialist will meet with caregiver at each clinic visit and provide information, education, disclosure skills, and support till disclosure occurs.
  Interventions: Behavioral: Disclosure intervention
- Usual care (Active Comparator): In the "enhanced usual care (control)" arm the disclosure specialist will meet with caregiver at each clinic visit and provide them will general health education and no mention or effort will be made to improve disclosure skills of caregiver.
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: Disclosure intervention — An adherence and disclosure specialist will meet with caregiver-child dyad at each clinic visit and provide caregiver information and skills for HIV disclosure till the caregiver discloses the HIV status to the child.
  Arms: Disclosure intervention
Behavioral: usual care — An adherence and disclosure specialist will meet with caregiver-child dyad at each clinic visit and provide caregiver with general health information without referencing HIV disclosure in their conversations till the caregiver discloses the HIV status to the child.
  Arms: Usual care

SUMMARY:
A culturally-relevant, theoretically and empirically sound, patient-centered, standardized disclosure intervention that can be integrated into routine clinical pediatric HIV care has potential to prevent transmission and improve the welfare of children and their caregivers in Ghana and other resource-limited settings. Results from this project will also further an understanding of factors and processes driving pediatric HIV disclosure.The study hypothesis is that several key barriers to disclosure of HIV status can be modified and the process of disclosure promoted with an intervention approach that is grounded in a traditional Ghanaian concept.

DETAILED DESCRIPTION:
The project aims to provide information on a structured disclosure intervention that can be integrated into usual care in Ghana and other resource-limited settings to improve the welfare of HIV-infected children and their caregivers. This area of investigation is profoundly understudied and of high importance to millions of children and their families in sub-Saharan Africa. While widely recognized as vital to better health outcomes, especially in the era of better access to HIV treatment, many children are not informed of their HIV diagnosis. A variety of sociocultural contextual barriers and deficient skills drive the persistent reluctance of caregivers and health care providers to inform children of the diagnosis. Our preliminary work shows that several key factors can be modified and the process of disclosure promoted with an intervention approach that is grounded in a traditional Ghanaian concept, "SANKOFA", and behavioral and bioecological systems theory. The patient-centered intervention approach uses an Adherence and Disclosure specialist model where a designated specialist familiar with the socio-cultural norms of the community is well trained to target modifiable information, motivation and behavioral skills of caregivers to facilitate their engagement in the process of disclosure (i.e., pre-disclosure, disclosure, and post-disclosure phases) in a manner suitable to the needs of the child.

The primary aims are: (1) To evaluate the effect of a structured, culturally-relevant disclosure intervention to caregivers delivered by a specialist as an integral component of routine HIV healthcare on the rate of caregiver disclosure of pediatric HIV at 1 year follow-up compared to treatment as usual, control condition, in a randomized trial and (2) To identify baseline characteristics (e.g., caregiver knowledge & motivation, child's age) predictive of caregiver disclosure of pediatric HIV independent of and in the presence of the structured disclosure intervention at 1 year follow-up.

Secondary aims are: (3) To assess whether the effect of HIV pediatric disclosure on medication adherence and health outcomes of children (virologic, immunologic, psychosocial, and behavioral) and the caregiver (psychosocial) varies by exposure vs non-exposure to the structured disclosure intervention and (4) To assess the fidelity and acceptability of the disclosure intervention over time among the clinic personnel designated disclosure specialist, caregiver, and children to whom HIV status has been disclosed. Provider, caregiver and child participants will be enrolled from tertiary HIV clinics in Ghana with longitudinal outcomes evaluated every 3 months post-randomization to 24 months post disclosure.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected children receiving care at the study sites
* started on antiretroviral therapy (ART) for the first time within 12 months of screening
* Or Child is going on ART at the time of screening
* Or child had achieved and maintained at least 25% of CD4+ T-lymphocytes according to age on treatment irrespective of duration of ART within 6 months prior to enrollment
* do not know their HIV diagnosis (based on caregiver account and medical records confirmation)

Exclusion Criteria:

* HIV-infected children less than 7 years
* HIV-infected children with congenital or developmental disorders
* HIV-infected children with comorbidities such as sickle cell disease or diabetes that require frequent clinic visits or hospitalizations
* Children with AIDS-defining illness or end stage AIDS.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 446 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
HIV disclosure rate | one year after intervention
  Structured and caregiver-centered and culturally-relevant disclosure intervention will be delivered by an adherence and disclosure specialist to the caregiver. After one year, the rate of disclosure of the HIV status of the children will be assessed.

SECONDARY OUTCOMES:
Baseline characteristics of caregiver predictive of disclosure to the child his/her HIV status | one year
  Baseline characteristics (e.g., caregiver knowledge & motivation, child's age) predictive of caregiver disclosure of pediatric HIV independent of and in the presence of the structured disclosure intervention at 1 year follow-up.
Medication adherence of children | two years
  The effect of HIV pediatric disclosure on medication adherence will be evaluated and compared between the two study arms - exposure vs non-exposure to the structured disclosure intervention.
Health outcomes of children | 2 years
  The effect of HIV pediatric disclosure on health outcomes of children (virologic - viral load, immunologic - CD4 count, psychosocial, and behavioral) will be evaluated and compared between the two study arms - exposure vs non-exposure to the structured disclosure intervention.
Health outcomes of caregiver | 2 years
  The effect of HIV pediatric disclosure on the psychosocial well being of the caregiver will be evaluated and compared between the two study arms - exposure vs non-exposure to the structured disclosure intervention.

OTHER OUTCOMES:
Fidelity of the disclosure intervention | 5 years
  The fidelity of the disclosure intervention over time among the clinic personnel designated disclosure specialist, caregiver, and children to whom HIV status has been disclosed will be assessed over the study period.
Acceptability of the disclosure intervention | 5 years
  The acceptability of the disclosure intervention over time among the clinic personnel designated disclosure specialist, caregiver, and children to whom HIV status has been disclosed will be assessed over the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Elijah Pantsil, MD, Principal Investigator — Yale University
Locations (2):
- Ghana (2):
  - Komfo Anoky Teaching Hospital, Kumasi, Ashanti Region
  - Korle-Bu Teaching Hospital, Accra, Greater Accra Region

REFERENCES:
- [Derived] Afrane AKA, Bobbala A, Martyn-Dickens C, Renner L, Antwi S, Kusah JT, Amissah K, Quaye D, Bosomtwe D, Gan G, Parziale S, Reynolds NR, Paintsil E, Shabanova V; Sankofa Study Team. Changes in caregiver psychosocial factors known to affect pediatric HIV disclosure: the Sankofa clinical trial experience in Ghana (2013-2023). AIDS Care. 2025 Dec 2:1-16. doi: 10.1080/09540121.2025.2594607. Online ahead of print. PMID 41330401
- [Derived] Shabanova V, Emuren L, Gan G, Antwi S, Renner L, Amissah K, Kusah JT, Lartey M, Reynolds NR, Paintsil E; Sankofa Study Team. Pediatric HIV Disclosure Intervention Improves Immunologic Outcome at 48 Weeks: The Sankofa Trial Experience. J Acquir Immune Defic Syndr. 2023 Dec 1;94(4):371-380. doi: 10.1097/QAI.0000000000003292. PMID 37643414
- [Derived] Radcliffe C, Sam A, Matos Q, Antwi S, Amissah K, Alhassan A, Ofori IP, Xu Y, Deng Y, Reynolds NR, Paintsil E; Sankofa Team. Sankofa pediatric HIV disclosure intervention did not worsen depression scores in children living with HIV and their caregivers in Ghana. BMC Public Health. 2020 Oct 20;20(1):1578. doi: 10.1186/s12889-020-09678-2. PMID 33081739
- [Derived] Farthing H, Reynolds NR, Antwi S, Alhassan A, Ofori IP, Renner L, Amissah KA, Kusah JT, Lartey M, Paintsil E; Sankofa Study Team. Illness Narratives of Children Living with HIV Who Do Not Know Their HIV Status in Ghana: I'm Sick, But I Don't Know the Sickness-A Qualitative Study. AIDS Behav. 2020 Nov;24(11):3225-3231. doi: 10.1007/s10461-020-02884-4. PMID 32333207
- [Derived] Paintsil E, Kyriakides TC, Antwi S, Renner L, Nichols JS, Amissah K, Kusah JT, Alhassan A, Ofori IP, Catlin AC, Gan G, Lartey M, Reynolds NR; Sankofa Study Team. Clinic-Based Pediatric Disclosure Intervention Trial Improves Pediatric HIV Status Disclosure in Ghana. J Acquir Immune Defic Syndr. 2020 May 1;84(1):122-131. doi: 10.1097/QAI.0000000000002316. PMID 32049772
- [Derived] Ofori-Atta A, Reynolds NR, Antwi S, Renner L, Nichols JS, Lartey M, Amissah K, Tettey JK, Alhassan A, Ofori IP, Catlin AC, Gan G, Kyriakides TC, Paintsil E; Sankofa Study Team. Prevalence and correlates of depression among caregivers of children living with HIV in Ghana: findings from the Sankofa pediatric disclosure study. AIDS Care. 2019 Mar;31(3):283-292. doi: 10.1080/09540121.2018.1537463. Epub 2018 Oct 25. PMID 30360643
- [Derived] Nichols JS, Kyriakides TC, Antwi S, Renner L, Lartey M, Seaneke OA, Obeng R, Catlin AC, Gan G, Reynolds NR, Paintsil E; Sankofa Study Team. High prevalence of non-adherence to antiretroviral therapy among undisclosed HIV-infected children in Ghana. AIDS Care. 2019 Jan;31(1):25-34. doi: 10.1080/09540121.2018.1524113. Epub 2018 Sep 20. PMID 30235940